CLINICAL TRIAL: NCT01232530
Title: Pharmacovigilance for Artemisinin-based Combination Treatments in Africa
Brief Title: Pharmacovigilance for ACTs in Africa
Acronym: PVACT
Status: Completed | Type: Observational
Sponsor: Centre Muraz (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Tinto Halidou, Theme leader of the Drug Resistance and alternative therapeutics, Centre Muraz
Other Study IDs: WHO/TDR - A70283
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Malaria
Keywords: Malria, ACT, Safety, Efficacy, pregarnancy
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood spot on filter paper for PCR analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Safety Active Surveillance Group: For the active surveillance, all age groups, including children less than 5 years of age, will be identified from the census database and encouraged to attend the health facility whenever sick. Those with a diagnosis of malaria and treated with an antimalarial drug will be actively monitored for AEs.
- Safety Passive Surveillance Group: For the people under passive surveillance, sick subjects attending the health facilities, diagnosed with malaria and treated with an antimalarial drug will be identified from the census database. The treatment administered will be recorded in a drug exposure log book and the patients will be encouraged to report passively any AE/ADR.
- Early Pregnancy Exposure to ACTs Group: All the pregnant women identified during the repeat surveys will be included in a pregnancy cohort. At the time the pregnant woman is identified, her possible exposure to ACTs will be extracted from the drug exposure log book or elicited by history. Births identified through the repeat surveys or any other outcome of pregnancy will be retrospectively matched with antimalarial treatment exposure, particularly during the first trimester of the pregnancy.
- ACT Effectiveness Monitoring Group: Besides monitoring AEs and ADRs, data on the effectiveness of ACTs when used in "real life" conditions and on a large scale will be collected in the active surveillance area. For patients with a microscopically confirmed diagnosis of malaria, clinical symptoms and a blood sample for thick and thin blood smears, will be collected before antimalarial treatment, at day 28 after treatment and at any unscheduled visit. Treatment administration will not be supervised.

SUMMARY:
This is a phase IV open label study assessing the safety and effectiveness of artemisinin derivatives-based combination therapy (ACT) when used on a large scale and under "real life" conditions.

DETAILED DESCRIPTION:
The study will be conducted in a well defined population in Burkina Faso by setting up a population-based monitoring system.

The monitoring for adverse events (AEs) will use two approaches (active and passive) based on a repeat survey of the study population. The active surveillance population will be weekly and actively visited at home at day 7, day 14 and day 28 after drug administration. The passive surveillance population will be encouraged to report passively any AE/ADR and they will NOT be actively visited at home.

In addition, the possible exposure to ACTs of all the pregnant women identified during the repeat surveys in both the active and passive surveillance areas will be extracted from the drug exposure log book or elicited by history, and the data will be entered into a pregnancy register.

For the effectiveness study, patients with a microscopically confirmed diagnosis of malaria (any parasite density), clinical symptoms and a blood sample for thick and thin blood smears, and later PCR analysis (on filter paper) for genotyping will be collected before antimalarial treatment, at day 28 after treatment and at any unscheduled visit. This will be repeated for each confirmed malaria episode.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females living in Nanoro DSS catchment area;
* Signed (or thumb-printed whenever patients are illiterate) informed consent.
* Patients' willingness and ability to comply with the study protocol for the duration of the study.

Exclusion Criteria:

* Severe malaria.
* Danger signs: not able to drink or breast-feed, vomiting (> twice in 24hours), recent history of convulsions (>1 in 24h), unconscious state, unable to sit or stand.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Initially, a census of the population living in Nanoro department and around (approximately 50,000 people) will be carried out. The complete census database will be utilized to estimate the incidence of malaria episodes and to determine whether there is any clustering of malaria episodes as well as AEs. Such census will be updated by a team of 8 field workers who will visit each single household every 4 months, for at least 3 years to identify newly pregnant women and to collect information on vital events such as births and deaths. Of the 50,000 people in the census database, approximately 25,000 will be under active surveillance while the other 25,000 will be under passive surveillance.
Sampling Method: Probability Sample
Enrollment: 3176 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Halidou Tinto, PharmD, PhD, Principal Investigator — Centre Muraz
Locations (1):
- Clinical Research Unit of Nanoro (CRUN) / Centre Muraz, Nanoro, Boulkiemdé, Burkina Faso

REFERENCES:
- [Derived] Sondo P, Bihoun B, Tahita MC, Derra K, Rouamba T, Nakanabo Diallo S, Kazienga A, Ilboudo H, Valea I, Tarnagda Z, Sorgho H, Lefevre T, Tinto H. Plasmodium falciparum gametocyte carriage in symptomatic patients shows significant association with genetically diverse infections, anaemia, and asexual stage density. Malar J. 2021 Jan 7;20(1):31. doi: 10.1186/s12936-020-03559-0. PMID 33413393
- [Derived] Sondo P, Derra K, Diallo Nakanabo S, Tarnagda Z, Kazienga A, Zampa O, Valea I, Sorgho H, Owusu-Dabo E, Ouedraogo JB, Guiguemde TR, Tinto H. Artesunate-Amodiaquine and Artemether-Lumefantrine Therapies and Selection of Pfcrt and Pfmdr1 Alleles in Nanoro, Burkina Faso. PLoS One. 2016 Mar 31;11(3):e0151565. doi: 10.1371/journal.pone.0151565. eCollection 2016. PMID 27031231
- [Derived] Tinto H, Sevene E, Dellicour S, Calip GS, d'Alessandro U, Macete E, Nakanabo-Diallo S, Kazienga A, Valea I, Sorgho H, Vala A, Augusto O, Ruperez M, Menendez C, Ouma P, Desai M, Ter Kuile F, Stergachis A. Assessment of the safety of antimalarial drug use during early pregnancy (ASAP): protocol for a multicenter prospective cohort study in Burkina Faso, Kenya and Mozambique. Reprod Health. 2015 Dec 4;12:112. doi: 10.1186/s12978-015-0101-0. PMID 26637464
- [Derived] Sondo P, Derra K, Diallo-Nakanabo S, Tarnagda Z, Zampa O, Kazienga A, Valea I, Sorgho H, Owusu-Dabo E, Ouedraogo JB, Guiguemde TR, Tinto H. Effectiveness and safety of artemether-lumefantrine versus artesunate-amodiaquine for unsupervised treatment of uncomplicated falciparum malaria in patients of all age groups in Nanoro, Burkina Faso: a randomized open label trial. Malar J. 2015 Aug 20;14:325. doi: 10.1186/s12936-015-0843-8. PMID 26289949